CLINICAL TRIAL: NCT05592522
Title: Is External Oblique Intercostal Block Under Enhanced Recovery After Bariatric Surgery (ERABS) Superior to Oblique Subcostal Transversus Abdominus Block? A Randomized Control Trial
Brief Title: Efficacy of External Oblique Intercostal Block in Laparoscopic Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al Mashfa Medical Center (Other)
Responsible Party: Principal Investigator, Dr. Mohamed Ibrahim Elsayed, Anesthesia consultant, Al Mashfa Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1/10-2022
Record Dates: First submitted 2022-10-19; First posted 2022-10-24 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Bariatric Surgery Candidate; Pain, Postoperative; Narcotic Use; Analgesia
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EOI group (Experimental): Ultrasound-guided bilateral external oblique intercostal (EOI) using 30 ml of 0.25% bupivacaine hydrochloride and oblique subcostal transverse abdominis plane (OSTAP) block using Placebo (NSS 0.9%) 30 ml combined with bilateral posterior rectus sheath block with 15 ml bupivacaine 0.25%.
  Interventions: Other: External oblique intercostal block; Other: Posterior Rectus sheath block
- OSTAP group (Experimental): Ultrasound-guided bilateral oblique subcostal transverse abdominis plane (OSTAP) block using 30 ml of 0.25% bupivacaine hydrochloride and external oblique intercostal (EOI) using Placebo (NSS 0.9%) 30 ml combined with bilateral posterior rectus sheath block with 15 ml bupivacaine 0.25%.
  Interventions: Other: Oblique subcostal TAP block; Other: Posterior Rectus sheath block

INTERVENTIONS:
Other: External oblique intercostal block — EOI block:Under guidance of the linear high frequency transducer, sagittal plane between anterior axillary line and midclavicular line at the level of the 6th rib, In-plane approach between external oblique and intercostal muscles Hydrodissection with 30 ml of 0.25% bupivacaine hydrochloride .
  Other Names: EOI
  Arms: EOI group
Other: Oblique subcostal TAP block — OSTAP block: The needle was inserted in plane through the rectus adjacent to costal margin Once the tip of the needle was visualized in between the rectus muscle and transversus abdominus muscle and negative pressure aspiration was demonstrated, 30 ml bupivacaine 0.25% was deposited within the plane and hydrodissection was noted.
  Other Names: OSTAP
  Arms: OSTAP group
Other: Posterior Rectus sheath block — Posterior rectus sheath block: Under linear ultrasound probe, the needle was advanced gradually through the rectus muscle posteriorly toward its medial edge, approaching the rectus sheath. After negative aspiration,12.5 mL bupivacaine 0.25% was injected until the rectus muscle was separated from the posterior rectus sheath by hydrodissection.
  Other Names: PRSB

SUMMARY:
Laparoscopic bariatric procedures nowadays are employed under ERAS protocol as an ambulatory surgery. Pain after laparoscopic procedures arises significantly from port site incisions in the anterior abdominal wall, and shoulder pain (referred from visceral pain). Narcotic medications are utilized to manage postoperative pain, but its disadvantages include, increased post-operative nausea and vomiting (PONV), ileus, sedation and delayed hospital discharge.

Oblique subcostal transversus abdominis plane block (OSTAP) had been studied before and found to be effective in reducing post-operative morphine usage and produce good analgesia for about 24hours postoperatively.

The ultrasound-guided external oblique intercostal (EOI) block is a new technique which proved to produce unilateral analgesia at thoracic dermatomes supplying the anterior and lateral aspects of the upper abdomen.

The aim of this study was to test the hypothesis that US-guided EOI blocks can produce more reduction in opioid usage during the first 24 h after of laparoscopic bariatric surgeries when compared to oblique subcostal TAP (OSTAP) block.

ELIGIBILITY:
Inclusion Criteria:

* age of 18 and 65;
* American Society of Anesthesia (ASA) class II or III
* elective laparoscopic bariatric procedure through trocars positioned at or above the um-bilicus (T10 dermatome).

Exclusion Criteria:

* preoperative chronic use or contraindication to opioid or NSAID
* allergy to bupivacaine
* local skin infection at the injection site of EOI or OSTAP blocks
* liver or renal insufficiency
* psychiatric, or neurological disease
* prior open abdominal surgery above T10 dermatome
* patients converted to open surgery; and patients expected to be subjected to more tissue trauma.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2022-10-26 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
24h equivalent oral morphine consumption | 24 hour
  Total pethidine consumption, calculated as an equivalent oral morphine dose, during the 24 hours,
Numerical rating scale (NRS) | 24 hours
  Numerical rating scale (NRS) in the PACU, and on arrival to the ward at 0 hours then at 2, 4, 6, 12, and 24 hours postoperatively(NRS) with 0 = no pain, to 100mm = the worst imaginable pain at the specified time.

SECONDARY OUTCOMES:
Quality of recovery 40 score(QoR-40) | 24 hours
  Quality of recovery 40 score at 24 hours.Twelve questions measured the comfort state; 9 questions measured the emotional state; 7 questions measured the psychological state; 5 questions measured the physical independence and 7 questions measured the level of pain. Each question received a score of 1 to 5 with a worst possible score of 40 and a best possible score of 200
AMBULATION TIME | 24 hours
  Time to first independent ambulation
Readiness for discharge | 24 hours
  time to readiness for discharge were measured according to the modified postoperative discharge scoring system (PADSS). Patients were considered eligible for discharge if they achieved a total score ≥ 9 on the condition that the vital signs parameter score was not less than 2, and none of the other five parameters scored a zero

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed I ElSayed, Principal Investigator — Al Mashfa Medical Center
Locations (1):
- Al Mashfa medical center, Khobar, Eastern Provence, Saudi Arabia